CLINICAL TRIAL: NCT05117879
Title: Comparison of R0 Resection Rate Between Cold Snare Polypectomy, Cold Endoscopic Mucosal Resection and Hot Endoscopic Mucosal Resection for 1-2 cm Colorectal Sessile Serrated Lesions: a Randomized Control Trial
Brief Title: R0 Resection Rate Between CSP, cEMR and hEMR for 1-2 cm Colorectal SSLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending physician, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202008004RINC
Record Dates: First submitted 2020-11-05; First posted 2021-11-11 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2020-12

CONDITIONS: Residual Disease
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: Three groups: Cold snaring polypectomy, Cold EMR and Hot EMR
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold snaring polypectomy (Other): The sessile serrated adenoma size between 10-20mm would be resected by cold snaring polypectomy
  Interventions: Procedure: Cold snaring polypectomy/ Cold EMR/Hot EMR
- Non-electrocautery Endoscopic Mucosal Resection (Cold EMR) (Other): The sessile serrated adenoma size between 10-20mm would be resected by cold EMR
  Interventions: Procedure: Cold snaring polypectomy/ Cold EMR/Hot EMR
- Electrocautery Endoscopic Mucosal Resection( Hot EMR) (Other): The sessile serrated adenoma size between 10-20mm would be resected by Hot EMR
  Interventions: Procedure: Cold snaring polypectomy/ Cold EMR/Hot EMR

INTERVENTIONS:
Procedure: Cold snaring polypectomy/ Cold EMR/Hot EMR — Cold snaring polypectomy: The technique of cold snare polypectomy is used to remove [small colonic polyps] without diathermy, which implies that a polyp is transected by a snare along with a rim of surrounding normal mucosa.
  Cold EMR: Cold EMR technique comprising submucosal injection of succinylated gelatin and dilute methylene blue before piecemeal cold snare resection of target polyp with a margin of normal tissue.
  Hot EMR: Hot EMR technique comprising submucosal injection of succinylated gelatin and dilute methylene blue before piecemeal electrocautery snare resection of target polyp with a margin of normal tissue.

SUMMARY:
Colorectal cancer is the most prevalent cancer and the third cancer related death in Taiwan. Adenoma is a precancerous lesion of colorectal cancer. Using colonoscopy to detect and remove the adenoma has a chance to prevent colorectal cancer development.

In the resection of colorectal polyps, for medium and large polyps that are more than one centimeter and less than two centimeters, because these polyps are at risk of cancer, they currently use hot-snaring polypectomy or more advanced endoscopic mucosal resection. Resection of such tumors ensures that a sufficient depth of resection and a high complete resection rate (R0 resection) are achieved.

Flat serrated adenoma (sessile serrated lesion) is a special adenoma that accounts for 10-12% of all colorectal polyps. Different from traditional adenomas, flat serrated adenomas within two centimeters in size have very little chance of becoming cancerous. And we know that on removal of medium and large polyps of 10-20mm, compared with the cold snaring polypectomy, the postoperative bleeding of the hot-snaring polypectomy technique is higher. Therefore, when removing low-risk polyps such as flat serrated adenomas, we may choose using a non-energized technique with low complications and we then would like to know whether the complete resection rate can be achieved by using the non-energized technique in the resection of a flat serrated adenoma of 10-20 mm, despite the large size, and compare the success rate and complications with traditional hot snaring polypectomy.

DETAILED DESCRIPTION:
This study is a single-country, multi-center, randomized controlled study. The subjects of the case were patients who underwent colonoscopy for various indications and found flat serrated adenomas ranging in size from 10-20 mm during the procedure. Excluded criterias are patients who are younger than 20 years old and have contraindications for colonoscopy. All patients included in the study will sign the informed consent sheet at the outpatient clinic. Once a flat serrated adenoma with a size of 10-20 mm is found during colonoscopy, the subjects will be randomly assigned to Cold snaring polypectomy group, cold endoscopic mucosal resection group or hot endoscopic mucosal resection group.

The preoperative preparation for bowel cleansing and colonoscope insertion method for these three groups of patients are totally the same as those of general colonoscopy. The only difference is the resection method flat serrated glands of 10-20 mm. The tumor was resected by cold snaring polypectomy, one group was resected by cold endoscopic mucosal resection, and the other group was resected by hot endoscopic mucosal resection. The endoscopists participating in this research project have extensive experience in endoscopy and perform at least one hundred polypectomy operations every year. The excised tumor will be sent to the pathology department for pathological diagnosis, and the pathology doctor will judge the completeness of the tumor resection

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 20 years old
2. Indicated for colonoscopy and willing to receive colonoscopy examination and polyp resection。
3. Any Sessile serrated adenoma size between 10-20mm was found during the examination。

Exclusion Criteria:

1. Age younger than 20 years old
2. Contraindication for colonoscopy or polypectomy (Such as recent acute myocardial infarction, pulmonary embolism ,coagulopathy..)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | within 14 days
  The margin of the resected specimen showed no adenoma involvement

SECONDARY OUTCOMES:
Mean polypectomy time | within 1 hour
  Total time spent for polypectomy and hemostasis technique
Successful tissue retrieval | 1 hour
  The rate of successful tissue retrieval after polypectomy
Mean number of cuts | 1 hour
  How many cuts to remove the lesion
En bloc resection | 1 hour
  The rate of en bloc resection
Cut number | 1 hour
  how many cuts to remove the lesion
Mean total procedure time | 1 hour
  The total time of the colonoscopy, including polypectomy or EMR
Emergency service visit | within 14 days
  Patient visit ER after polypectomy for any complication
Delayed bleeding rate | within 14 days
  Bleeding occurs delayed from several hours to weeks after the polypectomy
Perforation rate | two weeks
  perforation after polypectomy or EMR

CONTACTS AND LOCATIONS:
Overall Officials: Han-Mo Chiu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan (roc), Taiwan

IPD SHARING:
Plan to Share IPD: No